CLINICAL TRIAL: NCT03045640
Title: Adapting a Family Strengthening Intervention (FSI) to Improve Early Childhood Development (ECD) Outcomes
Brief Title: Family Strengthening Intervention for Early Childhood Development (ECD)
Acronym: FSIECD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: World Bank (Other)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15440_IVC
Record Dates: First submitted 2016-12-16; First posted 2017-02-07 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Child Development
Keywords: ECD; parenting program; home visiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FSI ECD (Experimental): Vulnerable Households (ubudehe 1 or 2) in the Government of Rwanda's poverty classification system, when categories ranged from 1 to 6; the system has since been restructured to have four categories only. Often a way to identify households for public works opportunities or other government assistance programs. For this arm, families had to be Ubudehe 1 or 2 and have a child aged 0-3 years. Households meeting these criteria in the catchment area(s) received the FSI ECD home-based parenting intervention from bachelor-level interventionists/"coaches."
  Interventions: Other: FSI ECD

INTERVENTIONS:
Other: FSI ECD — The FSI ECD intervention was delivered in a structured curriculum format, covering a range of topics from health, water and sanitation, good hygiene, early stimulation, conflict resolution, to good communication. It was designed to improve vulnerable households home environment and engagement with their children in order to improve child development outcomes. The curriculum was delivered by bachelor-level trained staff with beneficiaries on an individual, one on one basis, using active coaching to promote child well being and behaviors with caregivers.
  Other Names: Family Strengthening Intervention for ECD

SUMMARY:
Study activities were carried out to adapt and test a family-strengthening intervention to improve child development outcomes among families facing adversity in Rwanda.

DETAILED DESCRIPTION:
Qualitative research from past studies was used to adapt an existing family-strengthening intervention for HIV-AIDS affected families to extremely vulnerable families with children 0-3 in order to improve early childhood development outcomes. This small scale pilot was carried out to test the feasibility and acceptability of the intervention for extremely vulnerable families with young children in Rwanda.

In the first 10 families the intervention consisted of 21 modules, in the second iteration of the study with an additional 10 families, the curriculum was summarized into 15 modules. Modules were delivered by trained bachelor-level interventionists/home-visiting coaches and were delivered to families one on one in their respective homes. Modules were delivered on a weekly to biweekly basis and were flexible to the families needs and other responsibilities.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants must live in the study catchment area
* Caregiver(s) raising a child between 6 and 3 years old and Ubudehe 1 or 2 (Rwanda's poverty classification system)
* We will enroll both single and dual caregiver families to reflect population dynamics.
* Legal guardians may be aunts, uncles, grandparents, or foster parents

Exclusion Criteria:

* Potential participants that do not live in the study catchment area
* Do not have at least one child between the ages of 0 and 3 living in their household for whom they are the primary caregiver
* Are not classified as Ubudehe 1 or 2
* Have severe cognitive impairments which preclude their ability to speak to the research questions under study

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change: Ages and Stages Questionnaire | 12 months/18 months
  Child development

SECONDARY OUTCOMES:
Change: Hopkins Symptoms CheckList | 12 months/18 months
  Caregiver Mental Health
Change: MICS-5 | 12 months/18 months
  Water, Sanitation, and Hygeine
Change: Rwanda Comprehensive Food Security and Vulnerability Analysis and Nutrition Survey | 12 months/18 months
  Household Food Security
Change: Locally Derived Scale | 12 months/18 months
  Family Trust and Unity

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Betancourt, Sc.D, M.A., Principal Investigator — Boston College

REFERENCES:
- [Derived] Desrosiers A, Saran I, Albanese AM, Antonaccio CM, Neville SE, Esliker R, Jambai M, Feika M, Betancourt TS. Task-sharing to promote caregiver mental health, positive parenting practices, and violence prevention in vulnerable families in Sierra Leone: a pilot feasibility study. BMC Psychiatry. 2024 Nov 11;24(1):787. doi: 10.1186/s12888-024-06209-w. PMID 39529061